CLINICAL TRIAL: NCT06764082
Title: Nutritional Intervention With High Chain Triglyceride Formulation During Perioperative Period of Kasai Surgery for Biliary Atresia: a Prospective Multicenter Trial
Brief Title: Nutritional Intervention for Biliary Atresia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Feng Jiexiong, pediatric surgery department, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nutr-BA
Record Dates: First submitted 2025-01-03; First posted 2025-01-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Nutrition Disorder, Infant; Biliary Atresia
MeSH Terms: conditions — Infant Nutrition Disorders; Biliary Atresia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high MCT group (Experimental): At a high-calorie concentration, each 1000 mL could provide 800 kcal, 15.8 g MCT, and 21.5 g protein (osmotic pressure 227 mOsm/kg). On the basis of 130 - 150% DRI, a high-calorie formula feeding amount of 160 ml/kg/d could provide 2.7 g/kg/d MCT.
  Interventions: Dietary Supplement: high MCT formula
- normal treatment group (Active Comparator): The recommended energy input was 130-150% of the reference intake (DRI) based on age and gender as per WHO. The final dosage and schedule were determined by the children and their parents or caregivers.
  Interventions: Dietary Supplement: normal oral intake of the traditional formula

INTERVENTIONS:
Dietary Supplement: high MCT formula — Energy Intake: The tube-feeding formula was a special medical-purpose formula food with high MCT and deep hydrolyzed milk protein (Alfare, Nestlé, Switzerland), which contained hydrolyzed whey protein, maltodextrin, vegetable oil, and MCT, etc. At a high-calorie concentration, each 1000 mL could provide 800 kcal, 15.8 g MCT, and 21.5 g protein (osmotic pressure 227 mOsm/kg).
  Feeding Procedure: On the basis of 130 - 150% DRI, a high-calorie formula feeding amount of 160 ml/kg/d could provide 2.7 g/kg/d MCT. After the operation, starting from when oral nutrition was feasible, the amount gradually increased from the initial amount until the expected amount was reached, and this continued until 6 months after the operation. The difference between the estimated feeding amount and the actual feeding amount could be selectively supplemented with enteral nutrition (nasogastric tube).
  Arms: high MCT group
Dietary Supplement: normal oral intake of the traditional formula — For the children in the control group, there were no special restrictions before the operation. After they were able to have a normal diet postoperatively, they were encouraged to have a normal oral intake of the traditional formula. The recommended energy input for the formula was 130 - 150% of the reference intake (DRI) based on age and gender as per the World Health Organization (WHO). The final dosage and schedule were determined by the children and their parents or caregivers. The feeding route and the schedule for complementary feeding were the same as those in the experimental group.
  Arms: normal treatment group

SUMMARY:
Infants with biliary atresia (Biliary atresia, BA) have an increased risk of malnutrition due to insufficient dietary intake to maintain normal growth, impaired intestinal absorption, increased metabolic rate, and damage to some liver macronutrient metabolic pathways. The medium-chain triglyceride formula (MCT) in enteral nutrition has advantages: (1) It has a fast metabolism in the liver and possesses the advantage of being an innate energy source; (2) It can share metabolic pathways with some other fatty acids (DHA, EPA), and can promote the synthesis of phospholipids, etc. Therefore, EN containing the MCT formula is regarded as an important approach to alleviate growth retardation in BA children and improve the nutritional status of patients. This study aims to observe the effect of intensified enteral feeding with a high MCT formula during the perioperative period compared to traditional oral feeding on the prognosis of children with biliary atresia. The method adopted is a prospective, two-arm, open-label, multicenter, and interventional real-world study.

ELIGIBILITY:
Inclusion Criteria:

* Infants under 3 months old;
* Children clinically diagnosed with biliary atresia and in need of Kasai surgery;
* The patient themselves, legal representative or guardian have signed the informed consent form and are willing to actively cooperate with treatment and follow-up.

Exclusion Criteria:

* Low birth weight infants or very low birth weight infants;
* Complicated with life-threatening diseases of various organ systems;
* Complicated with other severe digestive tract malformations or other diseases that may interfere with the treatment of the patient or the patient's compliance;
* Patients who have participated in other clinical trials within the last month;
* Any other conditions that the researcher deems unsuitable for participation in this trial.

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
age by weight Z score | 6 months
  scores

SECONDARY OUTCOMES:
age by height Z score | 6 months
  scores

OTHER OUTCOMES:
age by BMI Z score | 6 months
  scores
Jaundice clearance rate | 6 months
  rate
The incidence of post-operative cholangitis | 6 months
  rate
length of hospital stay | 2 weeks
  number

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR